CLINICAL TRIAL: NCT03098693
Title: Dyadic-Based Diagnosis, Care, and Prevention for HIV Discordant Couples in Tanzania
Acronym: DDCP
Status: Completed | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Michael Sweat, Professor, Director, Division of Global and Community Health, Director of MUSC Center for Global Health, Medical University of South Carolina
Other Study IDs: R01MH106369-01 (NIH); R01MH106369 (NIH)
Record Dates: First submitted 2017-03-22; First posted 2017-04-04 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-01

CONDITIONS: HIV
Keywords: Serodiscordant; Pre-exposure Prophylaxis; Self-testing; Tanzania

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sero-discordant Couple Cohort: We will enroll and track a cohort of 60 serodiscordant couples (120 individuals). The HIV-positive couple members will be offered anti-retroviral therapy (ART) and the HIV-negative couple members will be offered pre-exposure prophylaxis (PrEP). We will monitor monthly clinic visits for the couple and will conduct in-depth behavioral surveys at baseline, 6-, 12-, and 18-months.
  Interventions: Behavioral: HIV Self-Testing; Behavioral: Immediate Access to ART for HIV infected couple members; Behavioral: Access to PrEP for HIV uninfected couple members

INTERVENTIONS:
Behavioral: HIV Self-Testing — Access to home-based HIV self-testing kits for stable couples.
Behavioral: Immediate Access to ART for HIV infected couple members — Immediate access to ART for HIV infected couple members (per current Tanzanian standard of care).
Behavioral: Access to PrEP for HIV uninfected couple members — Access to PrEP for HIV uninfected couple members.

SUMMARY:
This is a prospective observational study of couples in Kisarawe, Tanzania who will be provided an intervention that offers: (1) HIV self-testing kits and pre-test counseling provided at the household, (2) linkage to a counseling and referral center for those who test positive, (3) facilitated enrollment to care and treatment for couples with confirmed HIV infection; and (4) access to pre-exposure prophylaxis for the negative partner in a HIV sero-discordant couple. We will identify HIV sero-discordant couples through the HIV self-testing component, and through identifying discordant couples at the local HIV clinic. HIV sero-discordant couples (N=64 couples) will be administered a baseline, 6- ,12-, and 18-month survey, and the investigators will collect ongoing clinical data from each clinic visit. Biometric data (fingerprint) will be collected at enrollment, and all encounters with the counseling and referral center, and HIV treatment center, to allow linking of utilization of services with survey data.

DETAILED DESCRIPTION:
The investigators propose to conduct a prospective observational study of cohabitating couples aged 18 years and above in Kisarawe, Tanzania who will be provided: (1) distribution of HIV self-testing kits to cohabitating couples; (2) linkage to confirmatory HIV-testing & counseling for those who test HIV-positive; (3) facilitated enrollment to care and treatment for those couples with confirmed HIV infection; and (4) for HIV serodiscordant couples, access to PrEP for the HIV-negative partner. A baseline survey, and a follow-up survey approximately 2 weeks later and HIV test, will be administered to all couples involved in the self-testing phase of the study. A cohort of 60 to 70 HIV serodiscordant couples will receive a survey at baseline 6-, 12-, and 18-month survey, and the investigators will collect ongoing clinical data from each clinic visit. Biometric data (fingerprint) will be collected at study and intervention encounters to link utilization of services with survey data. The investigators will also enroll serodiscordant couples from patients already receiving care from the Kisarawe Care and Treatment Center (CTC).

The specific AIMS evaluate 4 key strategic goals, including:

1. HIV Self-Testing for Stable Couples: (a) assess the acceptability, safety, and factors associated with uptake of HIV self-testing; and (b) determine the proportion of clients testing positive for HIV via self-testing who engage in care.
2. Dyadic Engagement of Sero-Discordant Couples in Care & Prevention: (a) establish the proportion of sero-discordant couples who will enroll in HIV care as a dyad, (b) determine the effect of dyadic care enrollment on HIV care retention and ART adherence, and (c) assess reduction in risk of acquiring HIV infection for the negative partner.
3. Pre-Exposure Prophylaxis (PrEP): (a) establish the proportion and characteristics of HIV negative clients in a sero-discordant relationship who opt to take PrEP, (b) determine how engaging in ARV treatment by the positive partner affects PrEP utilization by the negative partner, and vice versa, and (c) Identify patterns and correlates of risk reduction strategies that couples in care utilize over time (abstinence, ARV for positive partner, PrEP for negative partner, condom use).
4. Operational: (a) determine Dyadic-based Diagnosis, Care, & Prevention (DDCP) program cost and economic efficiency, (b) compare DDCP to clinic-based and mobile VCT with regard to cost and efficiency for testing and linkage to care, and (c) assess the feasibility, acceptability, safety, and utility of using biometric data to track service utilization.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for participation in the self-testing cohort, each individual has to be:

1. age 18 years or older (and at least one member of the couple has to be aged 55 years or below),
2. live in the household regularly,
3. have no plans for moving from the area before the follow up period.

To be eligible for the prevention and care portion of the study, couples must be:

1. in an HIV sero-discordant relationship,
2. pregnant or breastfeeding women will be allowed to enroll in the study after counseling on the risks and benefits is provided,
3. HIV-negative women who are pregnant or breastfeeding will be allowed to take PrEP after counseling on the risks and benefits is provided.

Exclusion Criteria:

Couples will not be eligible for enrolled in the sero-discordant sub-cohort if:

1. the HIV-negative member has signs of advanced kidney disease (measured by serum creatinine),
2. the HIV-negative partner has Hepatitis B and markers of poor liver functioning (measured by alanine aminotransferase).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Cohabitating couples aged 18 to 55 years of age, residing in Kisarawe Town, Tanzania. Our cohort will be comprised of HIV sero-discordant couples.
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2017-11-21 (Actual); Primary Completion 2020-09-07 (Actual); Study Completion 2020-09-07 (Actual)

PRIMARY OUTCOMES:
Utilization of HIV Self-Test Kits | 2 weeks
  The proportion of eligible individuals who received an HIV self-test kit who successfully used the kit within two weeks of receiving the test kit.
Sharing of HIV Test Results with Primary Partner | 18 months
  The self-reported proportion of study participants who told their primary partner the results of the HIV test generated by the self-test kit.
Proportion of HIV Sero-discordant Couples who Engage in HIV Care Together | 18 months
  Proportion of HIV Sero-discordant Couples who Engage in HIV Care Together
Adherence to ART Among HIV Infected Members of Sero-discordant Couples | 18 months
  Self-reported proportion of doses of ART medication successfully taken on recommended schedule.
Retention in ART Care | 18 months
  Having ≥2 outpatient visits at least 3 months apart per year
Uptake of PrEP | 18 months
  Proportion of eligible HIV-uninfected cohort members who opt to take PrEP
Uptake of ARVs | 18 months
  Proportion of eligible HIV-infected cohort members who opt to take ART
Adherence to ART prescription refills among HIV infected members of sero-discordant couples | 18-Months
  Proportion of ART prescriptions successfully filled based on pharmacy records among HIV-infected members of sero-discordant couples.
HIV Viral Load | 18-months
  Copies per mL of HIV detected in blood sample.
Reduction in HIV-related Risk Behaviors | 18 months
  Self-reported number of sexual partners.
Reduction in sex with non-primary sex partners | 18-Months
  Any self-reported sex with non-primary sexual partner.
Reduction in sex acts | 18-months
  Self-reported number of vaginal and anal sex acts.
Reduction in unprotected sex | 18-months
  Self-reported proportion of vaginal and anal sex acts in which a condom was used.

SECONDARY OUTCOMES:
Program cost per client served | 18 months
  Program cost per client served

CONTACTS AND LOCATIONS:
Locations (1):
- Muhimbili University of Health and Allied Programs, Dar Es Salaam, Coast Region, Tanzania

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-26): https://cdn.clinicaltrials.gov/large-docs/93/NCT03098693/Prot_SAP_000.pdf